CLINICAL TRIAL: NCT03363191
Title: A Randomised, Double-blind, Parallel Group, Multicentre Study to Compare the Efficacy of Fluticasone Furoate/Vilanterol 100/25mcg Versus Fluticasone Furoate 100mcg on Asthma Control in Patients With Uncontrolled Asthma
Brief Title: The Efficacy of Fluticasone Furoate/Vilanterol Versus (vs) Fluticasone Furoate on Asthma
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn due to an internal decision.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206962
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: fluticasone furoate/vilanterol, efficacy, asthma, Chronic obstructive pulmonary disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol; Albuterol

STUDY DESIGN:
Intervention Model Description: Subjects will receive either fluticasone furoate/vilanterol 100/25 mcg or fluticasone furoate 100 mcg once daily in this parallel group study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects received Fluticasone Furoate/Vilanterol (Experimental): Subjects will receive fluticasone furoate/vilanterol 100/25 mcg inhalation powder via ELLIPTA dry powder inhaler (DPI) once daily for the 12 week treatment period. Subjects will receive salbutamol/albuterol as rescue medication on an as-needed basis.
  Interventions: Drug: Fluticasone Furoate/Vilanterol; Drug: Salbutamol/Albuterol
- Subjects received Fluticasone Furoate (Active Comparator): Subjects will receive fluticasone furoate 100 mcg inhalation powder via ELLIPTA DPI once daily for the 12 week treatment period. Subjects will receive salbutamol/albuterol as rescue medication on an as-needed basis.
  Interventions: Drug: Fluticasone Furoate; Drug: Salbutamol/Albuterol

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol — Fluticasone furoate/vilanterol will be supplied as inhalation powder in ELLIPTA DPI. It will contain 2 strips with 30 blisters per strip. First strip will contain fluticasone furoate 100 mcg dry white powder blended with lactose. Second strip will contain vilanterol 25 mcg dry white powder blended with lactose and magnesium stearate.
  Arms: Subjects received Fluticasone Furoate/Vilanterol
Drug: Fluticasone Furoate — Fluticasone furoate will be supplied as inhalation powder in ELLIPTA DPI. It will contain a single strip with 30 blisters, containing fluticasone furoate 100 mcg dry white powder blended with lactose.
  Arms: Subjects received Fluticasone Furoate
Drug: Salbutamol/Albuterol — Salbutamol/albuterol will be provided to subjects to use as rescue medication on an as-needed basis.

SUMMARY:
The objective of this study is to evaluate fluticasone furoate/vilanterol compared with fluticasone furoate alone in subjects with asthma that is uncontrolled on low to mid dose inhaled corticosteroid (ICS) or low dose ICS/ long acting beta agonist (LABA) combination. This is a phase IV, randomized, double-blind, parallel group, multicenter study evaluating fluticasone furoate/vilanterol 100/25 micrograms (mcg) and fluticasone furoate 100 mcg once daily, delivered as an inhalation powder using the ELLIPTA® device in subjects with uncontrolled asthma despite daily ICS or ICS/LABA therapy. The study will measure treatment response and asthma control using the Asthma Control Questionnaire-7 (ACQ-7) focusing on symptomatic control. In this study, proportion of subjects with an improvement in ACQ-7 score of >=0.5 at Week 12 compared to Baseline for the fluticasone furoate/vilanterol 100 mcg/25 mcg and fluticasone furoate100 mcg groups will be assessed. The total study duration for each subject will be 17 weeks including 4-week run in period, 12-week treatment period and 1-week follow up period. Approximately 1012 subjects will be randomized into the study. ELLIPTA is a registered trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Screening Inclusion Criteria

* Capable of giving signed informed consent.
* Male or female subjects aged >= 18 years of age at Screening (Visit 1). A female subject is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies; Not a woman of childbearing potential (WOCBP); A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for the duration of the study.
* A diagnosis of persistent asthma for at least 12 weeks prior to Screening (Visit 1).
* All subjects must be using an ICS with or without LABA for at least 12 Weeks prior to Visit 1. Two populations are eligible for enrolment: Subjects maintained on a stable ICS low to medium-dose fluticasone propionate 100 to 250 mcg twice daily or equivalent for at least 4 weeks prior to Visit 1; Subjects maintained on a stable dose of an ICS/LABA low-dose combination product (e.g., SERETIDE/ADVAIR 100/50 mcg twice daily or equivalent, via other combination products or via separate inhalers) for at least 4 weeks prior to Visit 1.
* Subjects must have a best pre-bronchodilator FEV1 of 50% - 80% of their predicted normal value. Predicted values will be based upon Global Lung Function Initiative (GLI) equations for spirometry reference values.
* Subjects must demonstrate >=12% and 200 milliliter reversibility of FEV1 within 10 to 40 minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol (or an equivalent nebulized treatment with albuterol/salbutamol solution) at Visit 1. Subjects that have documented reversibility meeting the criteria above within the last 6 months prior to Visit 1 (Screening) will be eligible and do not need to repeat the reversibility assessment at Visit 1 (Screening). Reversibility measurements, including historical reversibility, should follow/meet the recommendations of the American Thoracic Society (ATS)/ European Respiratory Society (ERS) Task force: Standardization of Lung Function Testing.
* All subjects must be able to replace their current short-acting bronchodilator (SABA), or other reliever strategy, with albuterol/salbutamol at Visit 1 (Screening), to be used only on an as-needed basis for the duration of the study. Each subject must be judged capable of withholding albuterol/salbutamol for at least 6 hours prior to performing spirometric evaluations.
* Subjects must be able to read and complete the questionnaire and electronic daily diary themselves.

Screening Exclusion Criteria

* Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years.
* An asthma exacerbation requiring systemic corticosteroids within 12 weeks prior to Visit 1. Any exacerbation requiring overnight hospitalization requiring additional treatment for asthma within 6 months prior to Visit 1.
* Current tobacco smoker or has a smoking history of >=10 pack-years (20 cigarettes/day for 10 years).
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* A subject must not have current evidence of: Atelectasis - segmental or larger; Bronchopulmonary dysplasia; Chronic bronchitis; Chronic obstructive pulmonary disease (COPD) current or past diagnosis including asthma/COPD overlap; Pneumonia; Pneumothorax; Interstitial lung disease or any evidence of concurrent respiratory disease other than asthma.
* A subject must not have any clinically significant, uncontrolled condition, or disease state that, in the opinion of the investigator, would put the safety of the participant at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* A subject must not have used any investigational drug within 30 days prior to Visit 1 or within five half-lives (t1/2) of the prior investigational study, whichever is longer of the two periods.
* Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy, or excipients used with fluticasone furoate/vilanterol 100/25 or fluticasone furoate 100 (i.e., drug, lactose or magnesium stearate).
* History of severe milk protein allergy.
* Administration of prescription or non-prescription medication that would significantly affect the course of asthma, or interact with study treatment.
* A subject must not be using or require the use of immunosuppressive medications during the study.
* A subject will not be eligible if he/she has any infirmity, disability, disease, or geographical location which seems likely (in the opinion of the investigator) to impair compliance with any aspect of this study protocol.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub investigator, study coordinator or an employee of the participating investigator.

Randomisation Inclusion Criteria

* Uncontrolled asthma (ACQ-7 >=1.5 at Visit 2).
* Demonstrated and reported in a daily diary on >=4 of the last 7 consecutive days of the run-in period (not including the date of randomisation): a score of >=1 on the day-time symptom scores and/or; a score of >=1 on the night-time asthma symptom scores and/or; albuterol/salbutamol use.
* Compliance is defined as completion of all questions/assessments, both morning and evening, on >=4 of the last 7 days during the run-in period. This does not include the items collected for the Asthma Daily Symptom Diary (ADSD).
* Compliance is defined as use of run-in medication on >=4 of the last 7 consecutive days of the run-in period (not including the date of randomisation) recorded in the electronic subject diary.

Randomisation Exclusion Criteria

* Positive urine pregnancy test at Visit 2.
* Use of any prohibited medications during the run-in period or at Visit 2.
* Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subjects asthma status or the participant's ability to participate in the study.
* Evidence of a severe exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-subject hospitalization or emergency department (ED) visit due to asthma that required systemic corticosteroids between Visits 1 and 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-07 (Estimated); Primary Completion 2019-05-29 (Estimated); Study Completion 2019-05-29 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with an improvement in ACQ-7 score of >= 0.5 at Week 12 compared to Baseline | Baseline and at Week 12
  The ACQ-7 consists of five questions about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze) in the previous week, along with one question on daily bronchodilator use in the previous week, and a measure of lung function (forced expiratory volume in 1 second [FEV1] % predicted). The response options for all these questions consist of a zero (no impairment) to six (total impairment) scale. The questions are equally weighted, and the ACQ-7 score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). A score >= 1.5 indicates asthma that is not well controlled, while a mean score of <= 0.75 indicates asthma that is well controlled, with a change of 0.5 defined as the minimal clinically important difference.

SECONDARY OUTCOMES:
Change from Baseline in the percentage of rescue-free daytime periods during the 12-week treatment period | Baseline and up to Week 12
  Subjects will be issued an electronic diary for use during the study. Subjects will record daytime asthma symptoms scores and the number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the daytime period. Symptoms and rescue use will be recorded between Visits 1 (Week-4) and 4 (Week 12), once in the evening (reporting daytime symptoms) before taking any rescue medication or ICS. Each evening, participants will record an asthma symptom score using the following scale: 1 = no symptoms during the day 2 = symptoms for one short period during the day 3 = symptoms for two or more short periods during the day 4 = symptoms for most of the day which did not affect my normal daily activities 5 = symptoms for most of the day which did affect my normal daily activities, 6 = symptoms so severe that I could not go to work or perform normal daily activities.
Change from Baseline in the percentage of rescue-free night time periods during the 12-week treatment period | Baseline and up to Week 12
  Subjects will be issued an electronic diary for use during the study. Subjects will record night time asthma symptoms scores and the number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the night time period. Symptoms and rescue use will be recorded twice a day between Visits 1 (Week-4) and 4 (Week 12), once in the morning (reporting night time symptoms) before taking any rescue medication or ICS. Each morning, subjects will record an asthma symptom score using the following scale: 1 = no symptoms during the night, 2 = symptoms causing me to wake once (or wake early), 3 = symptoms causing me to wake twice or more (including waking early), 4 = symptoms causing me to be awake for most of the night, and 5 = symptoms so severe that I did not sleep at all.
Change from Baseline in the percentage of symptom-free daytime periods during the 12-week treatment period | Baseline and up to Week 12
  Subjects will be issued an electronic diary for use during the study. Subjects will record daytime asthma symptoms scores and the number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the daytime period. Symptoms and rescue use will be recorded between Visits 1 (Week-4) and 4 (Week 12), once in the evening (reporting daytime symptoms) before taking any rescue medication or ICS.
Number of subjects with an ACQ-7 score <= 0.75 at Week 12 | Baseline and at Week 12
  The ACQ-7 consists of five questions about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze) in the previous week, along with one question on daily bronchodilator use in the previous week, and a measure of lung function (FEV1 % predicted). The response options for all these questions consist of a zero (no impairment) to six (total impairment) scale. The questions are equally weighted, and the ACQ-7 score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). A score >=1.5 indicates asthma that is not well-controlled, while a mean score of <= 0.75 indicates asthma that is well-controlled, with a change of 0.5 defined as the minimal clinically important difference.
Change from Baseline in the percentage of symptom-free night time periods during the 12-week treatment period | Baseline and up to Week 12
  Subjects will be issued an electronic diary for use during the study. Subjects will record night time asthma symptoms scores and the number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the night time periods. Symptoms and rescue use will be recorded between Visits 1 (Week-4) and 4 (Week 12), once in the morning (reporting night time symptoms) before taking any rescue medication or ICS.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline